CLINICAL TRIAL: NCT04146181
Title: A Phase II, Multicenter, Single-arm, Open-label Study of SCT-I10A in Patients With Recurrent/ Metastatic Head and Neck Squamous Cell Carcinoma Who Progressed on or After Platinum-based Chemotherapy
Brief Title: Safety and Efficacy of SCT-I10A in Head and Neck Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCT-I10A-B201
Record Dates: First submitted 2019-10-28; First posted 2019-10-31 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SCT-I10A (Experimental): SCT-I10A, 200 mg intravenous (IV) on Day 1 of each 3-week cycle.
  Interventions: Drug: PD-1

INTERVENTIONS:
Drug: PD-1 — SCT-I10A, 200 mg intravenous (IV) on Day 1 of each 3-week cycle.
  Other Names: SCT-I10A

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of SCT-I10A for Recurrent/ Metastatic Head and Neck Squamous cell Carcinoma who progressed on or after platinum-based chemotherapy

DETAILED DESCRIPTION:
This is an open label, single-arm and multicenter phase II study designed to evaluate Objective Response Rate (ORR) of SCT-I10A for Recurrent/ Metastatic Head and Neck Squamous cell Carcinoma who progressed on or after platinum-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in this clinical trial and sign an informed consent form;
2. Male or female, age ≥ 18 years old;
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
4. Has histologically- or cytologically-confirmed recurrent or metastatic (disseminated) head and neck squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, and larynx;
5. Is considered incurable by local therapies;
6. Have measurable disease based on RECIST1.1. tumor lesions, situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesion after 3 months of radiotherapy;
7. Have provided tissue for PD-L1 biomarker analysis
8. The estimated survival period is ≥ 3 months;
9. Patients who have been treated with platinum (cisplatin/carboplatin/nidaplatin) and have clear disease progression during treatment (at least 2 cycles) or after treatment (see RECIST version 1.1) or side effects Intolerance, and the minimum dose of platinum drugs must meet:

   Minimum dose of cisplatin: ≥60mg/m2 per cycle, or ≥120mg/m2 in 8 weeks; The minimum dose of carboplatin: AUC ≥ 4 / cycle, or total AUC ≥ 8 within 8 weeks.

   If cisplatin is converted to platinum, the platinum dosage can be calculated using the following formula: carboplatin 1AUC = cisplatin 15mg/m2; The minimum dose of nedaplatin: ≥80mg/m2 per cycle, or ≥160mg/m2 in 8 weeks; Note: Platinum drugs can be used as adjuvant therapy for postoperative patients (synchronous radiotherapy), for palliative chemotherapy in patients with advanced stage or in patients with recurrent and/or metastatic disease.
10. Laboratory inspection:

    Blood routine: neutrophils ≥1.5×l09/L, platelets≥75×109/L, hemoglobin≥80g/L; Liver function: alanine aminotransferase (ALT) and aspartate aminotransferase (AST), ALT and AST ≤ upper limit of normal value × 3 for liver metastasis, ALT and AST ≤ upper limit of normal value for liver metastases × 5; total bilirubin ( TBIL) ≤ upper limit of normal value × 1.5; Renal function: creatinine (Cr) ≤ normal upper limit × 1.5; Coagulation: Activated Partial Thromboplastin Time (aPTT), International Normalized Ratio (INR), Prothrombin Time (PT) ≤1.5xULN Echocardiogram: LVEF≥50%
11. Subjects should agree to use an adequate method of contraception starting with the first dose of study medication through 6 months after the last dose of study therapy. Female subjects of childbearing potential should have a negative blood pregnancy test within 7 days prior to receiving the first dose of study medication, and should be non-breastfeeding;

Exclusion Criteria:

1. Disease is suitable for local therapy administered with curative intent
2. Prior therapy with an anti-PD-1 or anti-PD1-L1 or -L2 therapy, or anti-CD137, or anti-CTLA-4 therapy
3. Diagnosed and/or treated additional malignancy within 5 years of randomization, with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin, and/or curatively-resected in situ cervical cancers;
4. NCI CTCAE v5.0 Grading of Peripheral Neuropathy≥2;
5. Active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previous treated brain metastases may participate provided they are stable for at least 2 weeks prior to the first dose of study medication, have no evidence of new or enlarging brain metastases, and are not using steroids for at least 14 days prior to trial treatment. Subjects with asymptomatic BM (without neurological symptoms, not using steroids, tumor lesions≤1.5cm) may participate in condition that the tumor lesion should be regularly evaluated using identical imaging modality for each assessment, either MRI or CT scans;
6. At the time of enrollment, patients still had ≥2 toxic side effects (except for hair loss, hearing loss, tinnitus, dry mouth or platinum-induced grade 2 neurotoxicity) caused by previous anti-tumor treatment;
7. Has known serious allergic reaction to study medication or any component of the product, and has known serious allergic reaction to other monoclonal antibodies (NCI CTCAE v5.0≥3);
8. Has received anti-tumor therapy, including chemotherapy, hormonal therapy, immunotherapy, radiotherapy, and etc. within 4 weeks of the first dose of treatment, except palliative radiotherapy for bone pain;
9. Has received any Chinese traditional medicine for anti-cancer purpose within 1 week of the first dose of treatment;
10. Has undergone important surgery within 4 weeks prior to first dose of treatment or has scheduled an important surgery during the study;
11. Has received immunosuppressive drugs during the study or within 2 weeks prior to first dose of treatment, except for the following situations:

    Intranasal, inhaled, topical corticosteroids (e.g. intra-articular injections); Physiological dose for systemic prednisolone (≤10mg/d or equivalent); Short-term administration (≤7days) of corticosteroids for prophylaxis or treatment against non-autoimmune allergic disease
12. Has known active, and/ or history of autoimmune disease (systemic lupus erythematous, rheumatoid arthritis, inflammatory bowel disease, AITD, multiple sclerosis, vasculitis, glomerulonephritis), and is likely to get a recurrence, or is at high-risk (organ-transplanted patients need immunotherapy), except those with stable type 1 DM after fixed dose of insulin administration , or those with autoimmune hypothyroidism only require HRT, or those with skin disorders that does not require systemic treatment (e.g. eczema, rash <10% BSA, psoriasis without symptoms around eyes)
13. Has known interstitial lung disease, such as interstitial pneumonia, pulmonary fibrosis, except asymptomatic drug-induced pneumonitis or radiation pneumonitis
14. Has a known history of HIV
15. Has known active Hepatitis B (e.g. HBsAg reactive) or Hepatitis C(e.g. HCV RNA [quantitative] is detected)
16. has uncontrolled active infections within 2 weeks before enrollment
17. Has received a live vaccine within 4 weeks prior to first dose of study treatment, except
18. Is with clinical symptoms, required clinical intervention or stable time less than 4 weeks of serous cavity effusion (such as pleural effusion and ascites);
19. Has severe conditions, including NYHA III heart failure, IHD, history of MI within 3 months prior to first dose of study treatment, poorly controlled DM (FBS≥10mmol/L) or poorly controlled hypertension (SBP≥160mmHg and/ or DBP≥100mmHg)
20. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
21. Is currently participating in other clinical trials, or has participated in a study of an investigational agent and received study therapy, or used an investigational device, any of whose end date is within 4 weeks prior to the first dose of study medication
22. has alcohol or drug addiction;
23. Subjects who are considered unsuitable for participating in this study for various reasons at the discretion of the investigator，such as inability to comply with study and/or follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2019-10-31 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
ORR | 1 year
  ORR is defined as proportion of patients achieving complete response (CR) or partial response (PR) according to RECIST v1.1 during trial treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Guangxi Medical University Affiliated Tumour Hospital, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No